CLINICAL TRIAL: NCT04390854
Title: Efficacy of Combined Blood Clot and Platelet Rich Fibrin Scaffolds in Regeneration of Necrotic Immature Permanent Teeth (A Randomized Controlled Clinical Trial)
Brief Title: Efficacy of Combined Blood Clot and Platelet Rich Fibrin Scaffolds in Regeneration of Necrotic Immature Permanent Teeth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Teaching Assistant of Dental Public Health and Statistician, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: blood clot/ PRF & regeneration
Record Dates: First submitted 2020-05-08; First posted 2020-05-18 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Pulp Necroses
Keywords: Regenerative endodontics; Open apex; Immature necrotic teeth
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The radiographic specialist and the statistician will be blinded to treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Induced blood clot scaffold (Active Comparator)
  Interventions: Biological: Blood clot scaffold
- Induced blood clot scaffold combined with Platelet rich fibrin (Experimental)
  Interventions: Biological: Blood clot scaffold combined with PRF

INTERVENTIONS:
Biological: Blood clot scaffold — Bleeding will be induced in the canal by passing a size 30 sterile K-file 3 mm beyond the apex with the goal of having the entire canal filled with blood to the level of the cemento-enamel junction. Bleeding will be stopped just below the cemento enamel junction.
  Biodentine will be placed approximately 3-4 mm below the cementoenamel junction.
  Arms: Induced blood clot scaffold
Biological: Blood clot scaffold combined with PRF — Platelet-rich fibrin will be prepared by drawing the patient blood into a 10mL test tube without the addition of an anticoagulant. To prevent the blood from coagulating after coming in contact with the glass tube, it will be centrifuged immediately using a table top centrifuge** at 400 g force for 12 minutes. Then platelet-rich fibrin membrane will be placed into the canal space to a level 3 mm below the cemento-enamel junction using hand plugger following the induction of apical bleeding by passing a number 30 sterile hand file 3 mm beyond the apex of the tooth. Biodentine cap will be placed over the platelet-rich fibrin scaffold.
  Arms: Induced blood clot scaffold combined with Platelet rich fibrin

SUMMARY:
The aim of the present study is to assess clinically and radio-graphically the regenerative potential of immature permanent teeth with necrotic pulp using blood clot and Platelet rich fibrin scaffolds.

DETAILED DESCRIPTION:
30 immature necrotic permanent teeth in patients will be allocated and divided into two groups. Group 1 will be treated by regenerative procedure using blood clot as a scaffold and Group 2 will be treated with regenerative procedures using combined blood clot and Platelet rich fibrin as a scaffold.

ELIGIBILITY:
Inclusion Criteria:

* Necrotic incisors with immature roots
* Pulp space not needed for post and core.
* The patient has to be free from any coagulation disorders, with normal platelets count.
* Good oral hygiene
* Cooperative patient

Exclusion Criteria:

* Internal or external root resorption.
* Root fracture and/or alveolar fracture.
* Previous root canal treatment.
* Medically compromised patients
* Uncooperative patient

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Subjective pain assessment | 1 month
  The patient will be asked about the presence of any pain or discomfort. Pain severity will be categorized as: no pain - mild pain - moderate pain - severe pain
Subjective pain assessment | 3 months
  The patient will be asked about the presence of any pain or discomfort. Pain severity will be categorized as: no pain - mild pain - moderate pain - severe pain
Subjective pain assessment | 6 months
  The patient will be asked about the presence of any pain or discomfort. Pain severity will be categorized as: no pain - mild pain - moderate pain - severe pain
Subjective pain assessment | 12 months
  The patient will be asked about the presence of any pain or discomfort. Pain severity will be categorized as: no pain - mild pain - moderate pain - severe pain
Assessment of pulp vitality | 1 month
  Pulp vitality will be assessed using thermal and electric pulp sensibility tests
Assessment of pulp vitality | 3 months
  Pulp vitality will be assessed using thermal and electric pulp sensibility tests
Assessment of pulp vitality | 6 months
  Pulp vitality will be assessed using thermal and electric pulp sensibility tests
Assessment of pulp vitality | 12 months
  Pulp vitality will be assessed using thermal and electric pulp sensibility tests
Assessment of root development | 1 month
  Continued root development will be assessed using cone beam computed tomography (CBCT) and compared with the contra-lateral healthy tooth
Assessment of root development | 3 months
  Continued root development will be assessed using cone beam computed tomography (CBCT) and compared with the contra-lateral healthy tooth
Assessment of root development | 6 months
  Continued root development will be assessed using cone beam computed tomography (CBCT) and compared with the contra-lateral healthy tooth
Assessment of root development | 12 months
  Continued root development will be assessed using cone beam computed tomography (CBCT) and compared with the contra-lateral healthy tooth
Assessment of the size of periapical radiolucency | 1 month
  Size of the lesion will be assessed using the periapical index score. The PAI provides an ordinal scale of 5 scores ranging from 1 (healthy) to 5 (severe periodontitis with exacerbating features).
Assessment of the size of periapical radiolucency | 1 month
  Size of the lesion will be assessed using Cone Beam Computed Tomography (CBCT).
Assessment of the size of periapical radiolucency | 3 months
  Size of the lesion will be assessed using the periapical index (PAI) score. The PAI provides an ordinal scale of 5 scores ranging from 1 (healthy) to 5 (severe periodontitis with exacerbating features).
Assessment of the size of periapical radiolucency | 3 months
  Size of the lesion will be assessed using Cone Beam Computed Tomography (CBCT).
Assessment of the size of periapical radiolucency | 6 months
  Size of the lesion will be assessed using the periapical index (PAI) score. The PAI provides an ordinal scale of 5 scores ranging from 1 (healthy) to 5 (severe periodontitis with exacerbating features).
Assessment of the size of periapical radiolucency | 6 months
  Size of the lesion will be assessed using Cone Beam Computed Tomography (CBCT).
Assessment of the size of periapical radiolucency | 12 months
  Size of the lesion will be assessed using the periapical index (PAI) score. The PAI provides an ordinal scale of 5 scores ranging from 1 (healthy) to 5 (severe periodontitis with exacerbating features).
Assessment of the size of periapical radiolucency | 12 months
  Size of the lesion will be assessed using Cone Beam Computed Tomography (CBCT).

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud MS Hassan, M.Sc, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Mohamed Ibrahim, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt; Sybel M Moussa, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt; Nihal A Lehita, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Bakhtiar H, Vatanpour M, Rayani A, Navi F, Asna-Ashari E, Ahmadi A, Jafarzadeh H. The plasma-rich in growth factor as a suitable matrix in regenerative endodontics: a case series. N Y State Dent J. 2014 Jun-Jul;80(4):49-53. PMID 25219066
- [Background] Keswani D, Pandey RK. Revascularization of an immature tooth with a necrotic pulp using platelet-rich fibrin: a case report. Int Endod J. 2013 Nov;46(11):1096-104. doi: 10.1111/iej.12107. Epub 2013 Apr 13. PMID 23581794
- [Background] Yassen GH, Eckert GJ, Platt JA. Effect of intracanal medicaments used in endodontic regeneration procedures on microhardness and chemical structure of dentin. Restor Dent Endod. 2015 May;40(2):104-12. doi: 10.5395/rde.2015.40.2.104. Epub 2014 Dec 24. PMID 25984471
- [Background] Yassen GH, Sabrah AH, Eckert GJ, Platt JA. Effect of different endodontic regeneration protocols on wettability, roughness, and chemical composition of surface dentin. J Endod. 2015 Jun;41(6):956-60. doi: 10.1016/j.joen.2015.02.023. Epub 2015 Mar 29. PMID 25823403
- [Background] Neha K, Kansal R, Garg P, Joshi R, Garg D, Grover HS. Management of immature teeth by dentin-pulp regeneration: a recent approach. Med Oral Patol Oral Cir Bucal. 2011 Nov 1;16(7):e997-1004. doi: 10.4317/medoral.17187. PMID 21743418
- [Background] Lovelace TW, Henry MA, Hargreaves KM, Diogenes A. Evaluation of the delivery of mesenchymal stem cells into the root canal space of necrotic immature teeth after clinical regenerative endodontic procedure. J Endod. 2011 Feb;37(2):133-8. doi: 10.1016/j.joen.2010.10.009. PMID 21238791
- [Background] Cotti E, Mereu M, Lusso D. Regenerative treatment of an immature, traumatized tooth with apical periodontitis: report of a case. J Endod. 2008 May;34(5):611-6. doi: 10.1016/j.joen.2008.02.029. PMID 18436046
- [Background] Cehreli ZC, Isbitiren B, Sara S, Erbas G. Regenerative endodontic treatment (revascularization) of immature necrotic molars medicated with calcium hydroxide: a case series. J Endod. 2011 Sep;37(9):1327-30. doi: 10.1016/j.joen.2011.05.033. Epub 2011 Jul 13. PMID 21846559
- [Background] Law AS. Considerations for regeneration procedures. J Endod. 2013 Mar;39(3 Suppl):S44-56. doi: 10.1016/j.joen.2012.11.019. PMID 23439044